CLINICAL TRIAL: NCT00988676
Title: The Effect of Bowel Preparation Status on the Polyp Missing Rate During Colonoscopy: Prospective Study Using Tandem Colonoscopic Evaluation
Brief Title: The Effect of Bowel Preparation Status on the Polyp Missing Rate
Status: Completed | Type: Observational
Sponsor: Konkuk University Hospital (Other)
Collaborators: Konkuk University Medical Center (Other); Konkuk University (Other)
Responsible Party: Sung Noh Hong, Konkuk University Medical Center; Konkuk University School of Medicine; Konkuk University
Other Study IDs: KUH1010135
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2009-10

CONDITIONS: Colorectal Polyps; Colonoscopy; Bowel Preparation; Polyp Missing Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- colonoscopy

SUMMARY:
High quality bowel cleaning preparation was most important prerequisites of a accurate colonoscopy, because even a small amount of residual fecal matter can obscure small polyps and increase unnecessary procedure time. Until now, several studies evaluated the impact of bowel preparation on the quality of colonoscopy using comparison of the polyp detection rate in patients with adequate bowel preparation status to that in patients with inadequate bowel preparation status during colonoscopy. However, there was no direct measurement the effect bowel preparation status on the polyp missing rate, the quality of colonoscopy, using tandem colonoscopic evaluation in prospective setting.

DETAILED DESCRIPTION:
1. Study flow

1. All patients perform Colonoscopy

   * record the polyp size, shape, location and number
   * record the factors affecting polyp missing rate

     * Patients' age / gender
     * Indication of colonoscopy
     * colonoscopist career
     * colonoscopy withdrawal time
     * bowel preparation status according to scale of U.S. Multi-Society Task Force on colorectal cancer, Aronchick's scale and Ottawa bowel preparation quality scale
2. the patients needed or wanted to 2nd stage colonoscopic polypectomy (2nd stage polypectomy was performed within 6 month)

   * record additionally detected polyp - size, shape, location and number

ELIGIBILITY:
Inclusion Criteria:

* The patients underwent colonoscopy and 2nd stage colonoscopic polypectomy at Konkuk University Medical Center

Exclusion Criteria:

* Colonoscopy was not reached the caecum
* The patients with 10 or more polyps (who suspected polyposis syndrome)
* Bowel preparation was inadequate when 2nd stage colonoscopic polypectomy
* The patients with inflammatory bowel disease or suspected inflammatory bowel disease
* The patients had a history of bowel resection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients underwent colonoscopy and 2nd stage colonoscopic polypectomy at Konkuk University Medical Center
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Noh Hong, M.D., Study Director — Konkuk University Medical Center; Konkuk University School of Medicine
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea